CLINICAL TRIAL: NCT03387241
Title: A Double Blind, Double Dummy, Randomised, Multicentre, Two Arm Parallel Group Study to Assess the Efficacy and Safety of FLUTIFORM® pMDI (2 Puffs Bid) vs Seretide® pMDI (2 Puffs Bid) in Subjects Aged ≥12 Years With Moderate to Severe Persistent, Reversible Asthma
Brief Title: Efficacy of FLUTIFORM ® vs Seretide® in Moderate to Severe Persistent Asthma in Subjects Aged ≥12 Years
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mundipharma (China) Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FLT13-CN-301
Record Dates: First submitted 2017-11-10; First posted 2018-01-02 (Actual); Last update posted 2019-04-29 (Actual); Status verified 2019-04

CONDITIONS: Asthma
Keywords: moderate; severe; persistent; reversible; Seretide; Flutiform
MeSH Terms: conditions — Asthma; Lymphoma, Follicular | interventions — fluticasone-formoterol; Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A double blind, double dummy, randomised, multicentre, two arm parallel design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fluticasone/ Formoterol (Flutiform) (Experimental): Dosage Form:2 puffs
  Unit Strength:
  Low dose: 50/5 µg Mid dose: 125/5 µg High dose 250/10 µg Dosing Frequency:BID Mode of Administration:Inhaled
  Interventions: Drug: Fluticasone/ Formoterol
- Fluticasone/ salmeterol (Seretide) (Active Comparator): Dosage Form:2 puffs
  Unit Strength:
  Low dose: 50/25 µg Mid dose: 125/25 µg High dose 250/25 µg Dosing Frequency:BID Mode of Administration:Inhaled
  Interventions: Drug: fluticasone/ salmeterol

INTERVENTIONS:
Drug: Fluticasone/ Formoterol — See above
  Other Names: FLUTIFORM® pMDI (2 puffs bid)
  Arms: Fluticasone/ Formoterol (Flutiform)
Drug: fluticasone/ salmeterol — See above
  Other Names: Seretide® pMDI (2 puffs bid)
  Arms: Fluticasone/ salmeterol (Seretide)

SUMMARY:
A double blind, double dummy, randomised, multicentre, two arm parallel group study to assess the efficacy and safety of FLUTIFORM® pMDI (2 puffs bid) vs Seretide® pMDI (2 puffs bid) in subjects aged ≥12 years with moderate to severe persistent, reversible asthma.

DETAILED DESCRIPTION:
The primary objective is to show non-inferiority in the efficacy of FLUTIFORM ® pMDI (2 puffs bid) versus Seretide® pMDI (2 puffs bid) based on the change from the pre-dose forced expiratory volume in the first second (FEV1) at baseline to 2 hours post-dose FEV1 at Week 12.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects at least aged ≥12 years old.
2. Known history of moderate to severe persistent, reversible asthma for ≥ 6 months prior to the Screening Visit characterized by inadequate asthma control on treatment with an ICS alone OR controlled asthma on treatment with an ICS-LABA combination.
3. Demonstrated a pre-dose FEV1 of ≥ 40% to ≤ 80% for predicted normal values during the Screening Visit (Visit 1) following appropriate withholding of asthma medications (if applicable).

   * No LABA use within 12 hours and/or no SABA use within 6 hours of the PFT.
   * No SAMA (e.g., ipratropium) use within 8 hours and/or no LAMA (e.g., tiotropium) use within 72 hours of the PFT.
   * No use of inhaled ICS-LABA combination asthma therapy within 12 hours of the PFT.
   * Inhaled corticosteroids are allowed on the day of screening.
   * Oral Aminophylline should be withheld for at least 24 hours prior to the PFT.
4. Documented FEV1 reversibility of ≥ 12% (plus ≥ 200ml if the subject is older than 18 years old) within last 12 months which could be accepted by the investigator, or during the screening phase or at Visit 2.
5. Demonstrated satisfactory technique in the use of the study medication.
6. Females of child bearing potential or less than one year post-menopausal must have a negative serum pregnancy test recorded at the screening visit and a negative urine pregnancy test result prior to the first dose of study medication, be non-lactating, and willing to use adequate and highly effective methods of contraception throughout the study. A highly effective method of birth control is defined as those which result in a low failure rate (i.e., less than 1% per year) when used consistently and correctly such as sterilisation, implants, injectables, combined oral contraceptives, some IUDs (Intrauterine Device, hormonal), sexual abstinence or vasectomised partner.
7. Willing and able to enter information in the diary and attend all study visits.
8. Willing and able to substitute study medication for their pre-study prescribed asthma medication for the duration of the study.
9. Written informed consent obtained, for <18 years old subjects, both parental consent and subjects assent are needed.

Besides The Inclusion/Exclusion Criteria Checking, Additional Randomisation Criteria Required Following Run-In Period:

1. Demonstrated a pre-dose FEV1 of ≥ 40% to ≤ 80% for predicted normal values at Randomisation Visit (Visit 3) following appropriate withholding of asthma medications (if applicable).
2. ACQ score at Visit 3 ≥ 1.0.
3. Subjects with a good compliance with treatment or patient dairy. The definition of good compliance is that the completeness of diary during the last 14 days of the run-in period is at least 80%. The compliance on diary completeness will be assessed from the aspects below and agreed by the investigator and study Medical Monitor:

   1. Diary info has been filled out on ≥80% of the days during the last 14 days before randomization (e.g., at least 11 days with diary filled completed out of the last 14 days prior to randomization).
   2. 80% main items including the study endpoints related ones have been filled out within the last 14 days prior to randomization.
   3. No other significant incompliance judged by the investigator that indicates the potential future incompliance for critical data collection during the study treatment period.

Exclusion Criteria:

1. The adolescent subjects (age ≥ 12 years to <18 years) who are on ICS alone at a dose >250μg bid fluticasone or equivalent OR ICS-LABA combination at a dose of Seretide > 250/50 μg bid or equivalent.
2. Near fatal or life-threatening (including intubation) asthma within the past year.
3. Chest X-ray at the Investigator's discretion from clinical perspective that reveals evidence of clinically significant abnormalities not believed to be due to asthma.
4. Hospitalization or an emergency visit for asthma within the 4 weeks before the screening visit or during the screening visit.
5. Use of systemic (injectable or oral) corticosteroid medication within 1 month of the Screening Visit.
6. Omalizumab use within the past 6 months prior to the Screening Visit.
7. Current evidence or known history of any clinically significant disease or abnormality including uncontrolled coronary artery disease, congestive heart failure, myocardial infarction, or cardiac dysrhythmia. 'Clinically significant' is defined as any disease that, in the opinion of the Investigator, would put the subject at risk through study participation, or which would affect the outcome of the study.
8. In the investigator's opinion a clinically significant upper or lower respiratory infection within 4 weeks prior to the Screening Visit.
9. Significant, non-reversible, active pulmonary disease (e.g., chronic obstructive pulmonary disease (COPD), cystic fibrosis, bronchiectasis, tuberculosis).
10. Subject has a smoking history equivalent to ≥ 10 pack years (i.e., at least 1 pack of 20 cigarettes /day for 10 years or 10 packs/day for 1 year, etc.) or significant history of exposure to biomass fuel combustion which may be considered a plausible contributory cause to the subject's obstructive lung disease.
11. Current smoking history within 12 months prior to the Screening Visit.
12. Current evidence or known history of alcohol and/or substance abuse within 12 months prior to the Screening Visit.
13. Subject has taken B-blocking agents, tricyclic antidepressants, monoamine oxidase inhibitors, astemizole (Hismanal), quinidine type antiarrhythmics, or potent CYP 3A4 inhibitors such as ketoconazole within the past week.
14. Current use of medications other than those allowed in the protocol that will have an effect on bronchospasm and/or pulmonary function.
15. Current evidence or known history of hypersensitivity or contraindications to the investigational products or components, including the history of paradoxical bronchospasm after inhalation therapy as immediate increase in wheezing and shortness of breath.
16. Subject has received an investigational drug within 30 days of the Screening Visit (12 weeks if an oral or injectable steroid).
17. Subject is currently participating in another clinical study or has already been randomized in this study.
18. Mental incapacity, unwillingness, or language barrier precluding adequate understanding, cooperation or any factors might block patients from protocol defined visits and may impact the patient diary completion at the Investigator's discretion.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2017-06-02 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2020-03-30 (Estimated)

PRIMARY OUTCOMES:
The primary efficacy endpoint is the change in pre dose Forced Expiratory Volume in one second (FEV1) from baseline to 2-hours post dose FEV1 at Week 12. | 12 weeks
  The change in pre-dose FEV1 from baseline to the 2-hours post dose FEV1 values at Week 12 will be analysed using a repeated measures ANCOVA model with fixed terms for treatment, baseline pre-dose FEV1, asthma severity, dose group, week and treatment by week interaction, and centre as a random effect. The statistical model will be used to calculate the treatment difference for the change in pre-dose FEV1 to 2 hours post-dose FEV1 at Week 12 (FLUTIFORM® - Seretide), corresponding 95% CI and p-value from the one-sided test for non-inferiority.

SECONDARY OUTCOMES:
The key secondary efficacy endpoint is the change in pre dose FEV1 from baseline to pre dose FEV1 at Week 12. | 12 weeks
  The change in pre dose FEV1 from baseline to the pre dose FEV1 values at Week 12 will be analysed using a repeated measures ANCOVA model with fixed terms for treatment, baseline pre dose FEV1, asthma severity, dose group, week and treatment by week interaction, and centre as a random effect. The statistical model will be used to calculate the treatment difference for the change in pre-dose FEV1 from baseline at Week 12 (FLUTIFORM® - Seretide), corresponding 95% CI and p-value from the test for non-inferiority. Non-inferiority will be concluded if the lower limit of the 95% CI is greater than or equal to -200ml.
The change in pre dose FEV1 from baseline to 2-hours post dose FEV1 at Week 2 and Week 6 | 2 weeks,6 weeks
  The change in pre-dose FEV1 from baseline to the 2-hours post dose FEV1 values at baseline (post-IMP), Week 2 and Week 6 will be analysed using a repeated measures ANCOVA model with fixed terms for treatment, baseline pre-dose FEV1, asthma severity, dose group, week and treatment by week interaction, and centre as a random effect. The statistical model will be used to calculate the treatment difference for the change in pre-dose FEV1 to 2 hours post-dose FEV1 at Week 2 and Week 6 (FLUTIFORM® - Seretide), corresponding 95% CI and p-value from the one-sided test for non-inferiority.
The change in pre dose FEV1 from baseline to pre dose FEV1 at Week 2 and Week 6 | 2 weeks,6 weeks
  The change in pre dose FEV1 from baseline to the pre dose FEV1 values at Week 2 and Week 6 will be analysed using a repeated measures ANCOVA model with fixed terms for treatment, baseline pre dose FEV1, asthma severity, dose group, week and treatment by week interaction, and centre as a random effect. The statistical model will be used to calculate the treatment difference for the change in pre-dose FEV1 from baseline at Week 2 and Week 6 (FLUTIFORM® - Seretide), corresponding 95% CI and p-value from the test for non-inferiority. Non-inferiority will be concluded if the lower limit of the 95% CI is greater than or equal to -200ml.
The number and percentage of subjects who discontinue due to lack of efficacy will be summarised for each treatment group | up to 12 weeks
  The Odds Ratio for Seretide versus Flutiform, corresponding 95% CI and p-value will be presented
Change from baseline in daily morning and evening peak expiratory flow rate (PEFR) at Week 2, 6 and 12 and on average during the 12 week treatment period. | 2 weeks, 6 weeks, 12 weeks
  Morning and evening PEFR data obtained from the last 7 days prior to each visit will further be averaged for each subject to get a mean value which corresponds to the respective scheduled visit. The calculated morning and evening PEFR values at baseline, Week 2, Week 6 and Week 12 and change from baseline at each time point will be summarized by treatment group as continuous data.
Change from baseline in other lung function parameters (PEFR) at Week 2, Week 6 and Week 12. | 2 weeks, 6 weeks, 12 weeks
  The other in-clinic lung function (PEFR) values assessed at each time-point (baseline, Week 2, Week 6, Week 12 and end of study), and the change from baseline to each post-baseline time-point will be summarised by treatment group as continuous data.
  These lung function values will be analysed using the same methodology applied to the primary and key secondary endpoint, for change in pre- and 2 hour post-dose lung function, respectively.
Change from baseline in other lung function parameters (FVC) at Week 2, Week 6 and Week 12. | 2 weeks, 6 weeks, 12 weeks
  The other in-clinic lung function (FVC) values assessed at each time-point (baseline, Week 2, Week 6, Week 12 and end of study), and the change from baseline to each post-baseline time-point will be summarised by treatment group as continuous data.
  These lung function values will be analysed using the same methodology applied to the primary and key secondary endpoint, for change in pre- and 2 hour post-dose lung function, respectively.
Change from baseline in other lung function parameters (FEF25-75) at Week 2, Week 6 and Week 12. | 2 weeks, 6 weeks, 12 weeks
  The other in-clinic lung function (FEF25-75) values assessed at each time-point (baseline, Week 2, Week 6, Week 12 and end of study), and the change from baseline to each post-baseline time-point will be summarised by treatment group as continuous data.
  These lung function values will be analysed using the same methodology applied to the primary and key secondary endpoint, for change in pre- and 2 hour post-dose lung function, respectively.
Change in asthma symptom scores from baseline at Week 2, 6, and 12 and on average during the 12 week treatment period. | 2 weeks, 6 weeks, 12 weeks
  Asthma symptom scores obtained from the last 7 days prior to each visit will further be averaged for each subject to get a mean value which corresponds to the respective scheduled visit. The calculated asthma symptom score values at baseline, Week 2, Week 6 and Week 12 and change from baseline at each time point will be summarized by treatment group as continuous data.
Change in sleep disturbance scores from baseline at Week 2, 6, and 12 and on average during the 12 week treatment period | 2 weeks, 6 weeks, 12 weeks
  Sleep disturbance scores obtained from the last 7 days prior to each visit will further be averaged for each subject to get a mean value which corresponds to the respective scheduled visit. The calculated sleep disturbance score values at baseline, Week 2, Week 6 and Week 12 and change from baseline at each time point will be summarized by treatment group as continuous data.
Change in percentage of asthma control days from baseline at Week 2, 6, and 12 and on average during the 12 week treatment period. | 2 weeks, 6 weeks, 12 weeks
  Asthma control days will be defined as an asthma symptom score of 0 (no symptoms), a sleep disturbance score of 0 (slept through the night) and no inhalations of rescue medication. Asthma control scores obtained from the last 7 days prior to each visit will further be averaged for each subject to get a mean value which corresponds to the respective scheduled visit. The calculated percentage of asthma control days at baseline, Week 2, Week 6 and Week 12 and change from baseline at each time point will be summarized by treatment group as continuous data.
Proportion of patients achieving well controlled asthma [ ACQ(Asthma Control Questionnaire) score ≤ 0.75 units] at Week 12. | 12 weeks
  The number and percentage of subjects achieving well controlled asthma (ACQ score ≤ 0.75 units) at Week 12 will be summarised by treatment group. The data will be analysed using logistic regression with fixed terms for treatment, baseline ACQ score, asthma severity, dose group and centre as a random effect. The Odds Ratio for Seretide versus Flutiform, corresponding 95% CI and p-value will be presented. Subjects with missing data at Week 12 will be considered as subjects not achieving well controlled asthma for the purpose of analysis.
Change in asthma control questionnaire (ACQ) score from baseline to Week 2 and Week 12. | 2 weeks,12 weeks
  The ACQ questionnaire at each time-point (baseline, Week 2, Week 12 and end of study) and the change from baseline to each post-baseline time-point will be summarised by treatment group as continuous data.
Proportion of subjects achieving a decrease from baseline to Week 12 in ACQ(Asthma Control Questionnaire) score ≥ 0.5 units. | 12 weeks
  The number and percentage of subjects achieving a decrease from baseline to week 12 of ≥ 0.5 ACQ units will be summarised by treatment group. The data will be analysed using logistic regression with fixed terms for treatment, baseline ACQ score, asthma severity, dose group and centre as a random effect. The Odds Ratio for Seretide versus Flutiform, corresponding 95% CI and p-value will be presented. Subjects with missing data at Week 12 will be considered as subjects without a decrease of ≥ 0.5 ACQ units for the purpose of analysis.
Change in average number of occasions of daily rescue medication (salbutamol) use from baseline during the 12 week treatment period.(salbutamol) will as assessed based on subject diaries records | 12 weeks
  The mean number of occasions per day will be calculated from the subject diaries for the 12 week treatment and baseline period. For the baseline value, data from the last 7 days prior to first IMP intake will be used.
  The mean number of occasions per day during baseline and the 12 week treatment period and the change from baseline during the treatment period will be summarized treatment group as continuous data.
Asthma exacerbations (incidence of subjects with at least one treatment emergent asthma exacerbation and time to first treatment emergent asthma exacerbation). | 12 weeks
  Asthma exacerbations will be analyzed using two different data sources:
  1. Based on exacerbations documented in the CRF by the investigator
  2. Programmatically derived from the diary data and relevant CRF pages Analyses on exacerbations documented by the investigator on the CRF will be considered the main analyses. Analyses on exacerbations obtained programmatically from the diary data will be considered as supportive analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Yu, Study Director — victoria.yu@mundipharma.com.cn
Locations (1):
- China-Japanese Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Oba Y, Anwer S, Maduke T, Patel T, Dias S. Effectiveness and tolerability of dual and triple combination inhaler therapies compared with each other and varying doses of inhaled corticosteroids in adolescents and adults with asthma: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2022 Dec 6;12(12):CD013799. doi: 10.1002/14651858.CD013799.pub2. PMID 36472162